CLINICAL TRIAL: NCT04481022
Title: Development of Clinical Prediction Rule for Classifying Females With Patellofemoral Pain Syndrome Who Respond to Proximal Control Exercises
Brief Title: Developmental of Clinical Prediction Rule for Females Responding to Proximal Control Exercises
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Alaa Eldin, Mr, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PFPS clinical prediction rule
Record Dates: First submitted 2020-07-17; First posted 2020-07-22 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Patellofemoral Pain Syndrome Clinical Prediction Rule
Keywords: clinical predicton rule; proximal control exercises

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group will receive proximal control exercises (Other)
  Interventions: Other: proximal control exercises

INTERVENTIONS:
Other: proximal control exercises — study investigates the effectiveness of proximal control exercises for patients with PFPS in improving pain and function. The findings of this systematic review are consistent with previous evidence reporting effectiveness of exercise for PFPS. In particular, there is consistent moderate to high quality evidence (three RCT, one CCT, three cohort studies, and one case series) that proximal interventions provide relief of pain and improved function in the short term, whereas the knee programs have variable effectiveness. Physical therapists should consider using proximal interventions for early stage treatment for PFPS (Peters et al., 2013).
  After 4 weeks of a combined knee and hip strengthening exercise program, sedentary females with PFPS had a greater reduction in pain during stair descent compared to the group who performed knee strengthening exercises only. Both groups also showed significant improvement in function and pain during stair ascent (Fakuda et al., 2010).

SUMMARY:
the aim of study is to investigate the effect of body mass index (BMI), age, duration of symptoms, pain severity and knee angle valgus on patient̕̕s response to proximal control exercises.

DETAILED DESCRIPTION:
Patellofemoral pain syndrome (PFPS) is recognized as one of the most common lower-extremity disorders encountered by orthopaedic physical therapists. Females were 2.23 times more likely to develop PFPS than males. Various authors have suggested that hip weakness may be an impairment associated with PFPS, because poor hip control may lead to abnormal lower extremity or patellofemoral motions. Clinical prediction rules (CPRs) are tools designed to improve decision making in clinical practice by assisting practitioners in making a particular diagnosis, establishing a prognosis, or matching patients to optimal interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 35 years.
* Anterior or retropatellar knee pain of non-traumatic origin that was greater than six weeks duration and provoked by at least two predefined activities (prolonged sitting or kneeling, squatting, jogging or running, hopping, jumping, or stair walking).
* Pain on palpation of the patellar facets, or with step down from a 15 cm step, or double leg squat.

Exclusion Criteria:

1. Concomitant injury or pathology of other knee structures.
2. Previous knee surgery.
3. patellofemoral instability (history of sublaxation or dislocation; positive apprehension test).
4. knee joint effusion.
5. Osgood-Schlatter's.
6. hip or lumbar spine pain (local or referred).
7. physiotherapy within previous year; prior foot orthoses treatment or use of anti inflammatories or corticosteroids.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-03 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
level of pain | baseline
  visual analogue scale 100-mm horizontal line anchored by word descriptors at each end by no the left and worst imaginable pain on the right
functional status | baseline
  Kujala questionnaire is a 13-items knee specific self-report questionnaire. It documents response to six activities thought to be associated specifically with anterior knee pain syndrome (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp, inability to bear weight through the affected limb, swelling, abnormal patellar movement, muscle atrophy and limitation of knee flexion. This questionnaire was used to ssess the individual's functional status and PFPS experienced during specific functional tasks.
Dynamic knee valgus 2d frontal plane projection angle | baseline
  2D frontal plane projection angle (FPPA) analysis to measure dynamic knee valgus. for 2D FPPA analysis, the centers of each of hip, knee and ankle joints will be determined using a standard tape measure, markers will be placed at the midpoint of the ankle malleoli for the center of the ankle joint, midpoint of the femoral condyles to approximate the center of the knee joint, and on the proximal thigh at the midpoint of the line from the anterior superior iliac spine to the knee joint center.

SECONDARY OUTCOMES:
isometric muscle power of hip abductor and external rotation | baseline
  Hand held dynamometer will be used to asses isomteric hip abductor and isometric hip external rotator power

REFERENCES:
- [Background] Robinson RL, Nee RJ. Analysis of hip strength in females seeking physical therapy treatment for unilateral patellofemoral pain syndrome. J Orthop Sports Phys Ther. 2007 May;37(5):232-8. doi: 10.2519/jospt.2007.2439. PMID 17549951
- [Background] Earl JE, Hoch AZ. A proximal strengthening program improves pain, function, and biomechanics in women with patellofemoral pain syndrome. Am J Sports Med. 2011 Jan;39(1):154-63. doi: 10.1177/0363546510379967. Epub 2010 Oct 7. PMID 20929936
- [Background] Lesher JD, Sutlive TG, Miller GA, Chine NJ, Garber MB, Wainner RS. Development of a clinical prediction rule for classifying patients with patellofemoral pain syndrome who respond to patellar taping. J Orthop Sports Phys Ther. 2006 Nov;36(11):854-66. doi: 10.2519/jospt.2006.2208. PMID 17154139